CLINICAL TRIAL: NCT01083524
Title: A Phase I, Open-Label, Two Centre Study to Evaluate Dichloroacetate(DCA) in Advanced Pulmonary Arterial Hypertension.
Brief Title: Dichloroacetate (DCA) for the Treatment of Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCA 20001
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Hypertension (Idiopathic, Familial or Anorexigen-associated)
Keywords: Pulmonary arterial hypertension; Pulmonary hypertension; Dichloroacetate; Dichloroacetate Sodium; DCA
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Dichloroacetate Sodium 3.0 mg/kg, BID
  Interventions: Drug: Dichloroacetate Sodium
- Group 2 (Experimental): Dichloroacetate Sodium 6.25 mg/kg, BID
  Interventions: Drug: Dichloroacetate Sodium
- Group 3 (Experimental): Dichloroacetate Sodium 12.5 mg po bid
  Interventions: Drug: Dichloroacetate Sodium

INTERVENTIONS:
Drug: Dichloroacetate Sodium — 3 mg po bid for 28 weeks
  Other Names: DCA
  Arms: Group 1
Drug: Dichloroacetate Sodium — 6.25 mg po bid
  Other Names: DCA
  Arms: Group 2
Drug: Dichloroacetate Sodium — 12.5 mg po bid
  Other Names: DCA
  Arms: Group 3

SUMMARY:
Hypothesis: The small molecule and metabolic modulator Dichloroacetate (DCA) is safe, tolerated as a potential therapy in patients with moderate or severe Pulmonary Arterial Hypertension (PAH).

This is a Phase I, two centre study in subjects with PAH WHO functional class III-IV whose symptoms have been clinically stable on their prescribed medical treatment (which includes endothelin and/or phosphodiesterase type 5 inhibitors) for 8 weeks prior to enrollment. Such patients will be given either DCA 3.0 mg/kg BID (group I), 6.25 mg/kg BID (group II) or 12.5 mg/kg BID (group III) as an additional treatment for 16 weeks. The design is open-label with the subjects acting as their own controls.

Primary endpoint is the safety and tolerability of DCA. Secondary end points include: a) functional capacity including a change in the 6 minute walk form baseline, b) change in pulmonary vascular resistance (measured by right heart catheterization), c) right ventricular volumes and mass (measured by MRI), d) NT-proBNP levels changed from baseline, e) change in FDG-glucose uptake in the lung and right ventricle (measured by PET) and f) change in quality of life indices.

15 evaluable patients in each site are expected to be included.

DETAILED DESCRIPTION:
The vascular remodeling in PAH is a state of apoptosis-resistance. As in cancer, a switch from the anti-apoptotic glycolytic metabolism towards the pro-apoptotic oxidative phosphorylation metabolism, has been shown to cause regression of vascular remodeling and PAH in several animal models. This has been achieved with the small molecular DCA, an inhibitor of the mitochondrial enzyme pyruvate dehydrogenase kinase.

DCA has been used in humans for over 30 years, mostly in the treatment of inherited mitochondrial disorders and is also currently being evaluated as a potential therapy in cancer.

This is a first-in-humans, Phase I, two centre study (University of Alberta and Imperial College) in subjects with advanced PAH, whose symptoms have been clinically stable on their prescribed medical treatment for 8 weeks prior to enrollment. These treatments include standard (eg diuretics, warfarin) or specific PAH therapies (eg endothelin or phosphodiesterase type 5 inhibitors). From the known metabolism of the drugs involved, no pharmacokinetic interaction is anticipated. In line with most safety and efficacy studies, the design is open-label with the subjects acting as their own controls.

Patients with PAH who have been stable on their current therapy for the preceding 2 months will be given either DCA 3.0 mg/kg BID (group I), 6.25 mg/kg BID (group II) or 12.5 mg/kg BID (group III) as an additional treatment for 16 weeks. Following the baseline visit, the patients will be followed every week for the first month, and then at weeks 6, 8 10, 12 and 16. In weeks 1, 3, 6 and 10, the patients' status will be assessed by telephone interview.

At all the other visits: medical history and physical examination will be performed. With the exception of week 2 (unless clinically indicated), this will be combined with routine hematology and biochemistry and an assessment of functional capacity (6 minute walk test). Serum lactate and NT-pro-BNP levels will be measured and PDH activity assay will be performed. Urine will be obtained for DCA metabolite studies.

At baseline and 16 weeks: A cardiac catheterization to assess change in pulmonary hemodynamics; a routine cardiac MR (RV mass/volumes, MR angiography); FDG-PET to examine for an effect on regional lung or RV glucose uptake.

If tolerated well, the subjects will continue with their medication and return for follow-up assessments at Weeks 20, 24 and 28. At each follow-up visit, a physical examination will be performed and functional capacity will be assessed (6 minute walk test). At the Week 28 visit a routine cardiac MR will also be performed. Enrollment will continue until 30 evaluable subjects (15 in each site) are included.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 years or older
2. Willing and able to complete informed consent form.
3. Documented diagnosis of PAH:

   * idiopathic, associated with anorexigens or familial;
   * mean pulmonary arterial pressure >25 mm Hg, pulmonary capillary wedge pressure =/< 15 mm Hg and pulmonary vascular resistance >240 dynes/sec/cm5 (measured by catheter).
4. Receiving stable doses for at least 2 months of one or more medications that are approved for treatment of PAH (endothelin receptor antagonists or phosphodiesterase type 5 inhibitors). Note: Anticoagulant therapy can be adjusted according to target INR and diuretic dose can be adjusted as required.
5. Modified World Health Organization(WHO) classification III-IV; stable for at least 8 weeks prior to enrollment.
6. 6MWD, as performed at screening or within three months (12 weeks) prior to screening, of ≥ 150 meters.
7. Expected survival of > 6 months.
8. ALT or AST levels < 3 times the upper limit of normal
9. Sexually active subjects must use an acceptable method of contraception while participating in the study, consisting of:

   1. Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner of female subject
   2. Oral contraceptives (either combined or progestogen only) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm. Women of child-bearing potential using an oral contraceptive in combination with a double-barrier method of contraception are required to continue to use this form of contraception for 6 weeks following discontinuation of study medication
   3. Double-barrier method of contraception consisting of spermicide with either condom or diaphragm
   4. IUD with documented failure rate of less than 1% per year
10. Females of childbearing potential must have negative pregnancy test at screening and be willing to have additional pregnancy tests during the study.

Exclusion Criteria:

1. Previous treatment with any formulation of DCA.
2. Known allergy or hypersensitivity to any excipient of DCA.
3. Clinically significant biochemical abnormality.
4. Clinical evidence of pre-existing neuropathy.
5. Use of investigational product or device within 30 days prior to dosing, or known requirement for any investigational agent prior to completion of all scheduled study assessments.
6. Known to be positive for human immunodeficiency virus (HIV).
7. Additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities, including bleeding disorders, arrhythmia, organ transplant, organ failure, current neoplasm, poorly controlled diabetes mellitus, and serious neurological disorders.
8. Blood results (performed within 14 days from study registration) as outlined below:

   * Absolute neutrophil count (ANC)<1500 cells/mm3.
   * Platelets<100,000 cells/mm3.
   * Hemoglobin <10 g/dl. (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10 g/dl is acceptable.)
   * S-Urea > 25 mg/dl
   * Creatinine clearance ≤ 30 ml
   * Bilirubin > 2.0 mg/dl
   * ALT >3 x normal range
   * AST >3 x normal range
9. Pregnant or lactating at screening, or planning to become pregnant (self or partner) at any time during study.
10. Contraindication to magnetic resonance imaging.
11. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of DCA in patients with pulmonary arterial hypertension. | December 2010

SECONDARY OUTCOMES:
The change in pulmonary vascular resistance from baseline at 16 weeks, measured by cardiac catheterization; | December 2010
Functional capacity: change from baseline in Functional Class and 6 min walk | December 2010
Changes in Right Ventricular size/function (measured by MRI), biomarkers (NT-proBNP), lung/RV metabolism (measured by FDG-PET) | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos D. Michelakis, MD, Principal Investigator — University of Alberta; Martin R Wilkins, MD, Principal Investigator — Imperial College London
Locations (2):
- University of Alberta Hospital, Edmonton, Alberta, Canada
- Imperial College, London, United Kingdom

REFERENCES:
- [Result] McMurtry MS, Bonnet S, Wu X, Dyck JR, Haromy A, Hashimoto K, Michelakis ED. Dichloroacetate prevents and reverses pulmonary hypertension by inducing pulmonary artery smooth muscle cell apoptosis. Circ Res. 2004 Oct 15;95(8):830-40. doi: 10.1161/01.RES.0000145360.16770.9f. Epub 2004 Sep 16. PMID 15375007